CLINICAL TRIAL: NCT04311151
Title: Impact of Self-visualization of Epileptic Seizures on Patients' Perception of the Disease and Risk Behavior (VICE)
Brief Title: Impact of Self-visualization of Epileptic Seizures on Patients' Perception of the Disease and Risk Behavior
Acronym: VICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Isabel Flores, Registered Nurse, Parc de Salut Mar
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CEIm-PSMAR 2016/6859/I
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Epilepsy; Epilepsy; Seizure; Risk Behavior; Risk-Taking
Keywords: epilepsy, Risk-Taking, risk behavior, seizure, visualization
MeSH Terms: conditions — Epilepsy; Risk-Taking; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self seizures visualization group (Experimental): Visualization of the own epileptic seizures occured during hospital admission.
  Interventions: Procedure: own seizures visualization
- usual management (No Intervention): Usual way management

INTERVENTIONS:
Procedure: own seizures visualization — At the hospital discharge, patients
  Arms: self seizures visualization group

SUMMARY:
In Spain, an estimated 690,000 persons have epilepsy, of whom 270,000 have active epilepsy (defined as those who have had a seizure in the last 5 years). It is estimated that 30% of patients diagnosed with epilepsy are drug-resistant. Patients with loss of consciousness or impaired awareness during seizures are at higher risk of injury due to accidents. To prevent such injuries, it is important that patients are sufficiently knowledgeable about their disease to allow them to avoid risk behavior.

In this project, we want to know if visualization of self seizures has an impact on the perception of the severity of the disease, as well as on the risky behavior habits.

DETAILED DESCRIPTION:
Design: Quasi-experimental study with a control group. Intervention group: standard of care and self-visualization of epileptic seizures. Control group: standard of care.

Main aims:

To determine whether self-visualization of seizures in patients with epilepsy modifies risk perception compared with patients not viewing their own seizures.

To determine whether viewing their seizures leads patients with epilepsy to plan changes in their risk behavior compared with patients not viewing their own seizures.

Design: Quasi-experimental study with a control group. Intervention group: standard of care and self-visualization of epileptic seizures. Control group: standard of care.

Sample size: Accepting an alpha risk of 0.05 and a beta risk lower than 0.2 on bilateral comparison, 50 participants will be needed in the intervention group and 25 in the control group to detect statistically significant differences between the proportion of patients showing behavioral change. It is expected that behavioral change will occur in 40% of the intervention group and 10% of the control group and that losses to follow-up will be 10%.

Variables: Sociodemographic, risk perception, intention to change behavior, perception of disease severity, quality of life, mood/depression, personality traits, anxiety.

Data collection: pre and post visualization of self seizures, and three months after discharge.

A descriptive analysis will be performed, with percentages and frequencies for qualitative variables and mean ± standard deviation (or median [range] depending on the normality of the distribution) for quantitative variables. Inferential analysis will be conducted with the chi-square test or nonparametric tests depending on the behavior of the variables obtained.

This project has been approved by the Clinical Research Ethics Committee of the hospital performing the study.

ELIGIBILITY:
Inclusion Criteria:

1. for the control group: patients aged 18 years or older admitted to the Epilepsy Unit of Hospital del Mar who voluntarily accept to participate in the study after prior psychological assessment.
2. for the control group: patients admitted to the Epilepsy Unit of Hospital Germans Tries who voluntarily accept to participate in the study.

Exclusion Criteria:

* Patients with no risk behavior according to the ad hoc questionnaire administered on admission.
* Cognitive impairment preventing adequate comprehension of the study.
* Vision-impaired patients and those with language barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
change from baseline patient's perception of the severity of his or her own disease | five minutes pre-visualization and five minutes post-visualization of self seizures, and three months later.
  self reported perceived severity of the disease through a visual analog scale (VAS).
change from patient's habits/risk behavior | five minutes pre-visualization and five minutes post -visualization of self seizures, and three months later
  conducted interview through several questions in the VICE questionnaire, related to intention of change risky behavior habits

SECONDARY OUTCOMES:
baseline quality of life | During the hospital admission (pre visualization of self seizures)
  measure of the quality of life specifically in patients with epilepsy, through the Quality of Life in Epilepsy Inventory-10(QUOLIE-10), validated spanish version. This inventory ranges from 10 to 50. The higher the score, the worse quality of life.
baseline severity of depressive symptoms | During the hospital admission (pre visualization of self seizures)
  self reported severity of depressive symptoms through the Beck Depression Inventory Second Edition (BDI-II), validated spanish version. This inventory ranges from 0 to 63. The higher the score, the highest severity of depressive symptoms.
anxiety trait and state | five minutes pre-visualization and five minutes post -visualization of self seizures
  self reported anxiety trait and state through the State-Trait Anxiety Inventory-STAI, validated spanish version. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
  This is a two part questionnaire. The state part will be reported five minutes pre and post visualization of self seizures, while the trait part will be reported only five minutes pre visualization.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Flores, Principal Investigator — Parc de Salut Mar

IPD SHARING:
Plan to Share IPD: No
Not considered, since the data processing will be done on an aggregate basis.

REFERENCES:
- [Result] Serrano-Castro PJ, Mauri-Llerda JA, Hernandez-Ramos FJ, Sanchez-Alvarez JC, Parejo-Carbonell B, Quiroga-Subirana P, Vazquez-Gutierrez F, Santos-Lasaosa S, Mendez-Lucena C, Redondo-Verge L, Tejero-Juste C, Morandeira-Rivas C, Sancho-Rieger J, Matias-Guiu J. Adult Prevalence of Epilepsy in Spain: EPIBERIA, a Population-Based Study. ScientificWorldJournal. 2015;2015:602710. doi: 10.1155/2015/602710. Epub 2015 Dec 10. PMID 26783554
- [Result] Herman S. Intractable epilepsy: relapsing, remitting, or progressive? Epilepsy Curr. 2010 Nov;10(6):146-8. doi: 10.1111/j.1535-7511.2010.01383.x. No abstract available. PMID 21157541
- [Result] Bradley PM, Lindsay B, Fleeman N. Care delivery and self management strategies for adults with epilepsy. Cochrane Database Syst Rev. 2016 Feb 4;2(2):CD006244. doi: 10.1002/14651858.CD006244.pub3. PMID 26842929